CLINICAL TRIAL: NCT04055077
Title: Influence of High-flow Nasal Oxygenation on Spontaneous Ventilation in Patients of Different Anesthesia Risk Class During Analgo-sedation for Vitrectomy, Randomized Controlled Trial
Brief Title: Influence of HFNO on Spontaneous Ventilation in Patients of Different ASA Risk During Analgo-sedation for Vitrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Split, School of Medicine (Other)
Collaborators: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Anita Vukovic, MD, specialist of anesthesiology, reanimatology and intensive care, University of Split, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8.1-19/188-1A
Record Dates: First submitted 2019-08-02; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Noninvasive Ventilation; Respiratory Insufficiency; Moderate Sedation; Hypoxia; Airway Management; Vitrectomy
Keywords: Noninvasive Ventilation; Airway management; Vitrectomy; Adult; Moderate Sedation; Hypoxia
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Intervention Model Description: Investigators plan to conduct prospective, parallel group, randomized controlled clinical trial.
  In total, 126 participants will be included in this trial. These participants are patients scheduled for analgo-sedation for vitrectomy.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Anesthesiologist who interviews and examines patients scheduled for PPV under analgo-sedation will enroll eligible participants and offer procedure explanation with possibility to sign uniformed written consent. Unique personal hospital admission number (UPHAN) will be assigned to all eligible participants. Participants will be randomized to control or intervention group by using random numbers generator. Anesthesiologist who implements anesthesia will receive nontransparent envelope with assigned intervention provided by independent investigator and will not decide which participant will receive LFNO or HFNO. However, attending anesthesiologist and participants will unavoidably be aware of type of oxygenation applied. Collected data are objective measures. Investigator who collects data after procedure will be unaware of study protocol and will enter data to formatted database. Participants' data will be noted under UPHAN. Outcome assessors will be unaware of intervention applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ASA I/LFNO (Active Comparator): Low-flow nasal oxygenation (LFNO) O2 flow 5L/min, FiO2 40%
  Interventions: Device: Low-flow nasal oxygenation (LFNO) ASA I
- ASA II/LFNO (Active Comparator): Low-flow nasal oxygenation (LFNO) O2 flow 5L/min, FiO2 40%
  Interventions: Device: Low-flow nasal oxygenation (LFNO) ASA II
- ASA III/LFNO (Active Comparator): Low-flow nasal oxygenation (LFNO) O2 flow 5L/min, FiO2 40%
  Interventions: Device: Low-flow nasal oxygenation (LFNO) ASA III
- ASA I/HFNO (Experimental): High Flow nasal oxygenation (HFNO) O2 flow 40L/min, FiO2 40%
  Interventions: Device: High-flow nasal oxygenation (HFNO) ASA I
- ASA II/HFNO (Experimental): High Flow nasal oxygenation (HFNO) O2 flow 40L/min, FiO2 40%
  Interventions: Device: High-flow nasal oxygenation (HFNO) ASAII
- ASA III/HFNO (Experimental): High Flow nasal oxygenation (HFNO) O2 flow 40L/min, FiO2 40%
  Interventions: Device: High-flow nasal oxygenation (HFNO) ASA III

INTERVENTIONS:
Device: Low-flow nasal oxygenation (LFNO) ASA I — Active comparator LFNO: O2 flow 5 L/min, FiO2 40%
  Arms: ASA I/LFNO
Device: Low-flow nasal oxygenation (LFNO) ASA II — Active comparator LFNO: O2 flow 5 L/min, FiO2 40%
  Arms: ASA II/LFNO
Device: Low-flow nasal oxygenation (LFNO) ASA III — Active comparator LFNO: O2 flow 5 L/min, FiO2 40%
  Arms: ASA III/LFNO
Device: High-flow nasal oxygenation (HFNO) ASA I — Experimental HFNO: O2 flow 40 L/min, FiO2 40%
  Arms: ASA I/HFNO
Device: High-flow nasal oxygenation (HFNO) ASAII — Experimental HFNO: O2 flow 40 L/min, FiO2 40%
  Arms: ASA II/HFNO
Device: High-flow nasal oxygenation (HFNO) ASA III — Experimental HFNO: O2 flow 40 L/min, FiO2 40%
  Arms: ASA III/HFNO

SUMMARY:
Pars plana vitrectomy is minimally invasive endoscopic procedure which is usually performed in moderate analgo-sedation given by anesthesiologist combined with topical anesthesia and retrobulbar or Subtenon block performed by surgeon. Intravenously applied anesthetics can often lead to slower breathing rate or cessation of breathing which introduces risk of low blood oxygen level despite careful adjustment of anesthetics' dose and application of standard low-flow nasal oxygenation (LFNO). Respiratory instability is often accompanied by circulatory instability manifested by disturbances of heart rate and blood pressure. LFNO provides maximally 40% inspired fraction of oxygen and can cause discomfort of a patient due to coldness and dryness of inspired gas.

On the other hand, high-flow nasal oxygenation (HFNO) can bring up to 100% of inspired oxygen fraction to patient, providing noninvasive pressure support of 3-7 cmH2O in patients' upper airway which ensures better oxygenation especially in higher anesthesia risk patients. Because of carrying warmed and humidified air/oxygen mixture via soft nasal cannula, HFNO is better tolerated by patients.

In this trial investigators will compare effect of HFNO to LFNO during intravenously applied standardized analgo-sedation given for vitrectomy in normal weight patients of low and high anesthesia risk.

Investigators hypothesize that normal weight patients of low and high anesthesia risk, whose breathing pattern is preserved, receiving HFNO vs. LFNO during standardized analgo-sedation for vitrectomy will be more respiratory and circulatory stable, preserving normal blood O2 and CO2 level, breathing pattern, heart rate and blood pressure.

DETAILED DESCRIPTION:
Pars plana vitrectomy (PPV) is minimally invasive micro-endoscopic surgery of posterior eye chamber. Most often patients receive combination of loco-regional anesthesia (topical anesthetic plus retrobulbar or Subtenon block), performed by a surgeon, and moderate analgo-sedation, performed by an anesthesiologist. Although applied intravenous anesthetics are short-acting, carefully titrated and continuously infused, anesthesia can lead to cessation of adequate spontaneous patients' breathing detected as bradypnoea, hypoxia and hypercapnia reflecting respiratory instability of patient. Respiratory instability is accompanied by circulatory one, reflected in heart rate and blood pressure deflections from baseline values. Usually, before, during and after analgo-sedation until patient is awaken, low-flow nasal oxygenation (LFNO) of 2-6 L/min O2 is applied through nasal catheter providing maximum inspiratory fraction of oxygen (FiO2) of 40%. Beside coldness and dryness of LFNO (therefore causing discomfort to patient), LFNO is often inadequate to prevent respiratory instability manifested as hypoxia and hypercapnia and subsequent circulatory disturbances.

Anesthesia risk is classified by American Society of Anesthesiologists Physical Status Classification System (ASA classification system) where patients of ASA class I anesthesia risk are generally healthy without systemic disease, patients deployed to ASA class II group have mild disease, having no functional impairment, higher risk ASA III patients have one or more significant organ function impairment.

High-flow nasal oxygenation (HFNO) delivers to patient high flow heated and humidified oxygen/air mixture (up to 70 L/min, up to 100% FiO2) using soft nasal cannula. HFNO produces 3-7 cmH2O of positive end-expiratory pressure therefore supporting patients breathing effort and providing apnoeic oxygenation, decreasing pharyngeal airway dead space and resistance. The patients find HFNO more comfortable as delivered gas is heated and humidified. HFNO is usually used for oxygenation of patients with predicted difficult oroendotrachial intubation prior to anesthesia, in process of awakening from anesthesia in postanesthesia care units and during process of weaning from mechanical respiratory support in intensive care units.

Goal of this trial is to compare effect of HFNO and LFNO on oxygenation maintenance during standardized procedure of intravenous analgo-sedation in normal weight ASA I, II and III risk class patients for elective PPV.

Investigators hypothesize that application of HFNO compared to LFNO in patients with preserved spontaneous breathing during procedural analgo-sedation for PPV contributes to maintaining adequate oxygenation, consequently adding to greater patients periprocedural respiratory and circulatory stability. Investigators expect that HFNO will provide reduced bradypnoea intervals (bradypnoea <12 breaths/min, FoB 1/min), longer maintenance of adequate oxygenation, shorter intervals of desaturation (peripheral blood oxygen saturation - SpO2≤92%), reducing hypercapnia (expiratory carbon-dioxide - expCO2≥45 mmHg) and less airway opening maneuvers performed by attending anesthesiologist (AOM). These will prevent partial respiratory insufficiency detected by low SpO2 accompanied by low or normal expiratory carbon-dioxide level (expCO2), and global respiratory insufficiency detected by decreased SpO2≤92% and increased expCO2≥45 mmHg.

Investigators plan to conduct prospective, parallel group, randomized controlled clinical trial. Trial will be managed according to principles of Declaration of Helsinki for scientific clinical research and will be planned and guided according to CONSORT guidelines (Consolidated Standards of Reporting Trials). The trial has been approved by Hospital's Ethic Committee.

The source of information are going to be 126 adult patients scheduled for PPV under analgo-sedation. Eligible participants will be interviewed and examined ambulatory by anesthesiologist, their ASA status, difficulty of airway management and body mass index (BMI) evaluated. After initial examination inclusive and exclusive criteria will be distinguished. Eligible participants who give voluntarily their written consent of participation will be included in this study. After that, participants will be assigned to equal ASA I, II and III risk class group. Each group will be randomized to intervention (HFNO) and control (LFNO) subgroup by computer random numbers generator. Randomization will be used until adequate number of participants in every subgroup is reached.

Interventions: intervention subgroups participants will be oxygenated via nasal cannula using high flow (40 L/min) of humidified and heated oxygen in air mixture (FiO2 40%). HFNO will be applied by oxygenator (AirVO™2, Fisher and Paykell, New Zealand, Technomedika, Croatia d.o.o.) during procedural analgo-sedation for PPV maintaining spontaneous breathing. In control subgroups, LFNO will be applied via nasal catheter (Bauerfeind d.o.o. Zagreb, Croatia) using standard low-flow oxygen (5 L/min, FiO2 40%). In both groups concentration of oxygen delivered depends on oxygen flow which is regulated by standard flow-regulator (flowmeter). Oxygen is delivered through pipelines from central hospital gas supply or from portable cylinder gas supply.

Anesthesia procedure will be uniformed for all participants. Integrated noninvasive monitoring of circulatory function (heart rate - EKG, intermittent mean arterial pressure - sphygmomanometer) will be set (Compact 7; Medical Econet GmbH, Germany). Respiratory vital functions: oxygenation (pulse oximeter), heart rate and expCO2 by using capnometer (Capnostream™35 Portable Respiratory Monitor, Medtronic, Belgium).

Every participant will have established intravenous infusion of 250 ml NaCl 0.9% via intravenous cannula regulated by continuous flow (Extension set/CONTROL-A-FLO Regulator 19 "Male Luer Lock Adapter", Baxter/Agmar d.o.o. United States of America/ Croatia).

Oxygenation (HFNO or LFNO) will be continuously administered before institution of analgo-sedation until patients' awakening. It will be started 3 minutes before analgo-sedation (preoxygenation), continued during analgo-sedation and procedure of PPV (perioperative oxygenation) and up to 5 minutes after PPV and until patient is awake (postprocedural oxygenation).

Induction of analgo-sedation will be instituted by droperidol 1.25 -2.5 mg bolus accompanied by continuous infusion of target remifentanyl concentration up to 0.05 mcg/kg/min. Intensity of sedation will be measured by Ramsay's sedation scale (RSS). Moderate sedation (RSS 4) is characterized by: purposeful response to verbal or tactile stimulation, no intervention required for airway patency maintenance, adequate spontaneous ventilation and sufficient cardiovascular function. Surgeon will apply topical local anesthetic on conjunctiva which is followed by regional anesthesia (Subtenon or retrobulbar block). Intravenous analgo-sedation will be administered via perfusor (B.Braun, Melsungen, Germany). Analgo-sedation will be discontinued immediately after end of PPV.

Control of nasopharyngeal airway is achieved by using oropharyngeal airway, if necessary. Oropharyngeal airway (Airway; Vigon-Medicpro d.o.o.) will be inserted after achieving moderate analgo-sedation and only if base of tongue is closing airway by dropping on posterior pharyngeal wall. Every manipulation of patients airway by anesthesiologist will be documented (insertion of airway, jaw thrust maneuver).

Measuring:

SpO2, expCO2, heart rate (fC) and respiratory rate (fD) will be measured continuously, and simultaneously continuously noted in 5 minutes intervals - T0=before oxygenation, T1=15 minutes after instituting LFNO or HFNO after beginning of analgo-sedation, T2=when patient is awake after oxygenation ends.

Noninvasive measurement SpO2 will be performed by indirect method using a pulse oximeter on the index finger of the left hand (Compact 7, Medical ECONET GmbH, Germany).

Blood pressure measuring and mean arterial pressure calculation will be repeated intermittently in 5 minutes intervals prior to-, during analgo-sedation and after patient is awaken. All measured parameters will be noted in identical intervals.

The data will be collected uniformly by three researchers: an anesthesiologist who interviews and examines patients ambulatory, an anesthesiologist designated for procedural analgo-sedation and an anesthesiologist who will collect the data after the completion of the analgo-sedation procedure.

The investigator in charge of the data collection will collect it from the pre-operative ambulatory list and the anesthesiologist list. The anesthesiology sheet will include all data from the trend table of the monitored vital parameters and from the simultaneously noted respiratory rate (fD) per minute and the expCO2.

The data will be collected through non-invasive measurements: peripheral blood oxygen saturation (SpO2), heart rate (fC), respiratory rate (fD), blood pressure (mean arterial pressure - MAP), carbon dioxide exhaled values before, in the stabilization and at the end of the analgo-sedation, i.e. 5 minutes after awakening of the patient.

A fourth researcher will be in charge of entering the collected data into the database. The statistician will analyze the data.

Basic data analyses will be performed by statistician. Sample size is determined by statistic computing web program: http://www.stat.ubc.ca/~rollin/stats/ssize used statistic test Inference for Proportions:Comparing Two Independent Samples. Assessment of sample size is computed for two independent samples with assumption of clinically significant difference in patients' oxygenation: ≤88 and ≥99%. Statistical significance of difference will be inferred with 5% α-error, 50% β-error and study power 0.80.calculated size of sample is: 21 participant pro subgroup (total of 126 participants).

Possible biases and confounding variables could be caused by hypothermia of the participant and by sphygmomanometer pressure on the same arm where peripheral oxygenation level is measured. These difficulties can be bypassed by: adjustment of room temperature where analgo-sedation for PPV is performed and blood pressure measuring cuff placed on right arm (pulse oximeter placed on left index-finger).

Any possible event that may occur during analgo-sedation that causes deviation from the study protocol will be the reason for exclusion of the subjects from the study and the PPV will be continued under anesthesia according to the rules of good clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* normal weight ASA patients of risk class I, II and III
* moderate intravenous analgo-sedation
* pars plana vitrectomy

Exclusion Criteria:

* Conventional vitrectomy
* Obese
* Diseases of peripheral blood vessels
* Hematological diseases
* Psychiatric diseases
* Sideropenic anaemia
* Patient's refusal
* Ongoing chemotherapy or irradiation
* Remifentanyl and Xomolix allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Maintaining oxygenation above the level of hypoxemia. Measure: peripheral blood saturation (SpO2) before application of LFNO or HFNO. | Time 0=before oxygenation
  Normal range >92% Acceptable deflection from normal values of peripheral blood saturation (SpO2) significant for hypoxemia is ≤92%, while all values above will be considered normal. SpO2 will be observed during procedure so that we can confirm or exclude differences connected with practical application of LFNO and HFNO.
Maintaining oxygenation above the level of hypoxemia. Measure: peripheral blood saturation (SpO2) 15 minutes after institution of LFNO or HFNO. | Time 1=15 minutes after institution of LFNO or HFNO
  Normal range >92% Acceptable deflection from normal values of peripheral blood saturation (SpO2) significant for hypoxemia is ≤92%, while all values above will be considered normal. SpO2 will be observed during procedure so that we can confirm or exclude differences connected with practical application of LFNO and HFNO.
Maintaining oxygenation above the level of hypoxemia. Measure: peripheral blood saturation (SpO2) 5 minutes after discontinuing analgo-sedation and oxygenation (LFNO and HFNO). | Time 2=5 minutes after discontinuing analgo-sedation and oxygenation (LFNO and HFNO)
  Normal range >92% Acceptable deflection from normal values of peripheral blood saturation (SpO2) significant for hypoxemia is ≤92%, while all values above will be considered normal. SpO2 will be observed during procedure so that we can confirm or exclude differences connected with practical application of LFNO and HFNO.

SECONDARY OUTCOMES:
Maintaining of expiratory efficiency of spontaneous breathing below hypercapnia value. Measure: expiratory level of CO2 (expCO2) before oxygenation by LFNO or HFNO. | Time 0=before oxygenation by LFNO or HFNO
  Normal range: 34 - 45 mmHg. Acceptable deflection from normal values significant for hypercapnia: expCO2 > 45 mmHg.
Maintaining of expiratory efficiency of spontaneous breathing below hypercapnia value. Measure: expiratory level of CO2 (expCO2) 15 minutes after institution of LFNO or HFNO. | Time 1=15 minutes after institution of LFNO or HFNO
  Normal range: 34 - 45 mmHg. Acceptable deflection from normal values significant for hypercapnia: expCO2 > 45 mmHg.
Maintaining of expiratory efficiency of spontaneous breathing below hypercapnia value. Measure: expiratory level of CO2 (expCO2) 5 minutes after discontinuing analgo-sedation and oxygenation (LFNO or HFNO). | Time 2=5 minutes after discontinuing analgo-sedation and oxygenation (LFNO or HFNO).
  Normal range: 34 - 45 mmHg. Acceptable deflection from normal values significant for hypercapnia: expCO2 > 45 mmHg.
Maintaining of normopnoea and spontaneous ventilation: frequency of breathing. Measure: frequency of breathing before oxygenation by LFNO or HFNO. | Time 0=before oxygenation by LFNO or HFNO.
  Frequency of breathing. Normal range: 12-20 breaths per minute. Frequency of breathing (FoB) - number of breaths per minute.
Maintaining of normopnoea and spontaneous ventilation: frequency of breathing. Measure: frequency of breathing 15 minutes after institution of LFNO or HFNO. | Time 1=15 minutes after institution of LFNO or HFNO.
  Frequency of breathing. Normal range: 12-20 breaths per minute. Frequency of breathing (FoB) - number of breaths per minute.
Maintaining of normopnoea and spontaneous ventilation: frequency of breathing. Measure: frequency of breathing 5 minutes after discontinuing analgo-sedation and oxygenation (LFNO or HFNO). | Time 2=5 minutes after discontinuing analgo-sedation and oxygenation (LFNO or HFNO).
  Frequency of breathing. Normal range: 12-20 breaths per minute. Frequency of breathing (FoB) - number of breaths per minute.
Maintaining of normopnoea and spontaneous ventilation: frequency of bradypnoea during analgo-sedation and oxygenation by LFNO or HFNO (fBRP/min). | From the beginning of analgo-sedation and oxygenation by LFNO or HFNO up to 5 minutes after discontinuing analgo-sedation and oxygenation by LFNO or HFNO.
  Frequency of breathing. Normal range: 12-20 breaths per minute. Bradypnoea will be noted when number of breaths is less then 12 breaths per minute. Normal range: up to one episode of bradypnoea during procedure. Acceptable deflection from normal range: >1 episode of bradypnoea during procedure.
Maintaining of normopnoea and spontaneous ventilation: frequency of desaturation during time of analgo-sedation and oxygenation by LFNO or HFNO. | From the beginning of analgo-sedation and oxygenation by LFNO or HFNO up to 5 minutes after discontinuing analgo-sedation and oxygenation by LFNO or HFNO.
  Frequency of desaturation during time of analgo-sedation: fDE, SpO2<92%. Normal range fDE = 1/60 min. Acceptable deflection from normal range: a ratio higher than 1/60 min.
Maintaining of normopnoea and spontaneous ventilation: Duration of desaturation (DE/min) from the start until the end of analgo-sedation and oxygenation by LFNO or HFNO. | From the beginning of analgo-sedation and oxygenation by LFNO or HFNO up to 5 minutes after discontinuing analgo-sedation and oxygenation by LFNO or HFNO.
  Normal range: SpO2<92% up to one minute. Duration of desaturation longer than one minute will be considered as insufficient ventilation.
Measurement of procedural parameters: duration of analgo-sedation. | From the start of continuous sedative infusion up to 1 minute after discontinuing infusion of sedative.
  Duration of analgo-sedation (min) - expected duration (minutes).
Measurement of procedural parameters: duration of awakening. | Up to 5 minutes from the discontinuing infusion of sedative until patient is oriented and cooperative (RSS Score 2).
  Time to full awakening (min) - expected duration up to 5 minutes (minutes).
  Analgo-sedation intensity is objectively measured by "Six Points Ramsay Sedation Scale" (RSS) where:
  RSS score 1 indicates that patient is agitated and restless, RSS score 2 - patient is oriented and cooperative, RSS score 3 - patient is responding to commands only, RSS score 4 - patient is briskly responding to light glabellar tap, RSS score 5 - patient is sluggishly responding to light glabellar tap, RSS score 6 - patient is not responding.
Circulatory stability: heart rate before oxygenation by LFNO or HFNO | Time 0=before oxygenation by LFNO or HFNO
  Heart rate (HR/min): normal range 60-100/min. Acceptable deflection from normal values is <60/heartbeats/min significant for bradycardia, while all values up to 100 heartbeats per minute will be considered normal.
Circulatory stability: heart rate 15 minutes after institution of LFNO or HFNO. | Time 1=15 minutes after institution of LFNO or HFNO.
  Heart rate (HR/min): normal range 60-100/min. Acceptable deflection from normal values is <60/heartbeats/min significant for bradycardia, while all values up to 100 heartbeats per minute will be considered normal.
Circulatory stability: heart rate 5 minutes after discontinuing analgo-sedation and oxygenation (LFNO or HFNO). | Time 2=5 minutes after discontinuing analgo-sedation and oxygenation (LFNO or HFNO).
  Heart rate (HR/min): normal range 60-100/min. Acceptable deflection from normal values is <60/heartbeats/min significant for bradycardia, while all values up to 100 heartbeats per minute will be considered normal.
Circulatory stability: mean arterial pressure before oxygenation by LFNO or HFNO | Time 0=before oxygenation by LFNO or HFNO.
  Mean arterial pressure (MAP): normal range: 65 - 110/min Acceptable deflection from normal values is <65 mmHg significant for hypotension, >110 mmHg for hypertension.
Circulatory stability: mean arterial pressure 15 minutes after institution of LFNO or HFNO | Time 1=15 minutes after institution of LFNO or HFNO.
  Mean arterial pressure (MAP): normal range: 65 - 110/min Acceptable deflection from normal values is <65 mmHg significant for hypotension, >110 mmHg for hypertension.
Circulatory stability: mean arterial pressure 5 minutes after discontinuing analgo-sedation and oxygenation (LFNO or HFNO). | Time 2=5 minutes after discontinuing analgo-sedation and oxygenation (LFNO or HFNO).
  Mean arterial pressure (MAP): normal range: 65 - 110/min Acceptable deflection from normal values is <65 mmHg significant for hypotension, >110 mmHg for hypertension.

CONTACTS AND LOCATIONS:
Locations (1):
- University clinical hospital centre Zagreb, Croatia, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta S, Blinder KJ, Shah GK, Grand MG. Pars plana vitrectomy versus combined pars plana vitrectomy and scleral buckle for primary repair of rhegmatogenous retinal detachment. Can J Ophthalmol. 2011 Jun;46(3):237-41. doi: 10.1016/j.jcjo.2011.05.003. Epub 2011 May 27. PMID 21784208
- [Background] Becker DE, Haas DA. Management of complications during moderate and deep sedation: respiratory and cardiovascular considerations. Anesth Prog. 2007 Summer;54(2):59-68; quiz 69. doi: 10.2344/0003-3006(2007)54[59:MOCDMA]2.0.CO;2. PMID 17579505
- [Background] Frat JP, Goudet V, Girault C. [High flow, humidified-reheated oxygen therapy: a new oxygenation technique for adults]. Rev Mal Respir. 2013 Oct;30(8):627-43. doi: 10.1016/j.rmr.2013.04.016. Epub 2013 May 29. French. PMID 24182650
- [Background] Booth AWG, Vidhani K, Lee PK, Thomsett CM. SponTaneous Respiration using IntraVEnous anaesthesia and Hi-flow nasal oxygen (STRIVE Hi) maintains oxygenation and airway patency during management of the obstructed airway: an observational study. Br J Anaesth. 2017 Mar 1;118(3):444-451. doi: 10.1093/bja/aew468. PMID 28203745
- [Background] Nagata K, Morimoto T, Fujimoto D, Otoshi T, Nakagawa A, Otsuka K, Seo R, Atsumi T, Tomii K. Efficacy of High-Flow Nasal Cannula Therapy in Acute Hypoxemic Respiratory Failure: Decreased Use of Mechanical Ventilation. Respir Care. 2015 Oct;60(10):1390-6. doi: 10.4187/respcare.04026. Epub 2015 Jun 23. PMID 26106206
- [Background] Ni YN, Luo J, Yu H, Liu D, Ni Z, Cheng J, Liang BM, Liang ZA. Can High-flow Nasal Cannula Reduce the Rate of Endotracheal Intubation in Adult Patients With Acute Respiratory Failure Compared With Conventional Oxygen Therapy and Noninvasive Positive Pressure Ventilation?: A Systematic Review and Meta-analysis. Chest. 2017 Apr;151(4):764-775. doi: 10.1016/j.chest.2017.01.004. Epub 2017 Jan 13. PMID 28089816
- [Background] Morris K. Revising the Declaration of Helsinki. Lancet. 2013 Jun 1;381(9881):1889-90. doi: 10.1016/s0140-6736(13)60951-4. No abstract available. PMID 23734387
- [Background] Moher D, Schulz KF, Altman DG; CONSORT Group. The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. Clin Oral Investig. 2003 Mar;7(1):2-7. doi: 10.1007/s00784-002-0188-x. Epub 2003 Jan 31. PMID 12673431
- See also: American Society of Anesthesiologists (ASA). ASA physical status classification system 2014 Oct [internet]. schaumburg, Illinois, USA: ASA;2014. — https://www.asahq.org/standards-and-guidelines/asa-physical-status-classification-system
- See also: Interactive Statistical Pages [internet]. USA: Statpages.net;c2019 [cited 2019 Aug1] — http://statpages.info/
- See also: Programiz [internet]. Kupandole, Nepal: Parewa Labs Pvt. Ltd [cited 2019 Aug 1]. Flowchart in programming. — http://www.programmiz.com/article/flowchart-programming